CLINICAL TRIAL: NCT02198950
Title: Combined Determination of sTREM-1, PCT and CD64 in Diagnosing Sepsis: a Prospective, Bicentric Study
Brief Title: Combined Determination of sTREM-1, PCT and CD64 in Diagnosing Sepsis
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Gibot Sébastien, Prof, Central Hospital, Nancy, France
Other Study IDs: 2009-A00870-57
Record Dates: First submitted 2010-09-23; First posted 2014-07-24 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Critically Ill Patients
Keywords: sepsis; diagnosis; biomarker
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasmas
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: all patients admitted into the ICU

SUMMARY:
The purpose of this study is to determine wether the combined measurement of the soluble form of TREM-1, PCT and the determination of neutrophils CD64 expression could diagnose sepsis in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients admitted into the ICU

Exclusion Criteria:

* absence of social protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient admitted into the ICU
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of sTREM-1, PCT, and CD64, taken alone or in combination in diagnosing sepsis in ICU patients as defined by the expert panel | 28 days
  A prospective study will be conducted in 300 patients admitted to a medical Intensive Care Unit, assaying serum concentrations of soluble Triggering Receptor Expressed on Myeloid cells-1 (sTREM-1) and procalcitonin (PCT), and measuring the expression of the high affinity immunoglobulin-Fc fragment receptor I (FcγRI) CD64 on neutrophils (PMN CD64 index) in flow cytometry. These biomarkers will be tested for their association with the diagnosis of infection. The final diagnosis of infection will be done by independent experts blinded for the results of CD64, sTREM-1, and PCT results. A "Bioscore" combining these biomarkers will be constructed and validated in an independent prospective cohort from another center.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Gibot, MD, PhD, Study Chair — Central Hospital, Nancy, France
Locations (2):
- France (2):
  - Bocage Hospital, Dijon
  - Central hospital, Nancy